CLINICAL TRIAL: NCT02926534
Title: A Cross-sectional Study of the Socio-demographic and Other Determinants of Chronic Obstructive Pulmonary Disease (COPD) Among Those Who Smoke, Quit Smoking and Never-smoking Cigarettes
Brief Title: Cross-Sectional Study of COPD Prevalence Among Smokers, Ex-smokers and Never-Smokers in Almaty, Kazakhstan
Status: Completed | Type: Observational
Sponsor: Kazakhstan Academy of Preventive Medicine (Other)
Collaborators: Philip Morris International (Industry); Synergy Research Group (Industry); HealthCity LLP (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIS.PMI.2016.001
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease; smoking; prevalence; cross-sectional study; Kazakhstan
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Smokers: Individuals (men and women) between the ages of 35 and 59 (inclusive) who are currently smoking conventional cigarettes with a minimum of 10 pack-year smoking history
- Ex-smokers: Individuals (men and women) between the ages of 35 and 59 (inclusive) with a minimum of 10 pack-year smoking history who stopped smoking cigarettes between 1 and 5 years ago
- Never-smokers: Individuals (men and women) between the ages of 35 and 59 (inclusive) who are current non-smokers and with no history of smoking (control group)

SUMMARY:
The purpose of this study is to assess the prevalence of COPD among individuals aged 35 - 59 years based results of spirometry before and after bronchodilator, presence of structural changes in lungs (emphysema, inflammatory changes and thickening of the walls of the large and small airways)detected by computer tomography as well as the symptoms of COPD. The study has three study groups: smokers of conventional cigarettes; those who had quit smoking 1 - 5 years ago, and those who haven't smoked cigarettes.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death worldwide. An estimated 0.5 million individuals in Kazakhstan may be affected by COPD, and the number of affected individuals and of deaths from COPD are expected to increase as the population ages. A better understanding of the epidemiology, causes, and social and other determinants of the disease is needed in order to develop effective treatments and prevention strategies.

Although COPD is traditionally defined by airflow obstruction in a spirometry test, smoking-associated effects on the lungs related to COPD also include emphysema, gas trapping, and chronic bronchitis. Symptoms such as productive cough, dyspnea, and exercise intolerance may be dismissed as normal aging, especially in older former smokers. Information is sparse about effects of smoking on individuals not diagnosed as having COPD (based on spirometry), and data from high-resolution computed tomography (CT) scanning in these individuals are limited.

COPD is strongly associated with smoking, but not all smokers will develop COPD. Cigarette smoking continues to be a common addiction in Kazakhstan despite efforts to reduce its prevalence. The study objectives are to assess true prevalence of COPD based on pulmonary function assessment and structural changes (emphysema and large and small airway inflammation with thickening) identified by high-resolution computer tomography (CT-scan) in addition to standard spirometric criteria and symptoms of dyspnea, exercise limitations, and chronic bronchitis. Such comprehensive approach will allow for objective comparisons of (1) current smokers of conventional cigarettes - 500 participants, (2) those subjects who quit smoking within the past 1 - 5 years - 200 participants, and (3) those subjects who never smoked cigarettes - 200 participants.

Using high resolution CT in addition to spirometry and other types of lung function assessment will help to determine COPD prevalence among non-smokers, smokers of conventional cigarettes and those who quit smoking. COPD prevalence will be defined based on abnormal respiratory function assessed by standard spirometric tests and by using COPD assessment test (CAT) questionnaire, 6-minute walk test and a high-resolution computed tomographic (HRCT) scan of the chest of those patients with preserved pulmonary functions but with clinical symptoms.

The cross-sectional study is retrospective in a sense, as it will allow to collect historical data on smoking, smoking cessation, address socio-demographic and other differentials of smoking. The investigators will also address the relationship of liver disease with COPD. This will be determined based on presence of hepatitis B and C tests (antigens and antibodies), liver enzyme levels and concentration of alpha-1-antitripsine, which is related to the development of COPD. Current or former smokers who had a concomitant diagnosis of asthma will not be excluded in the cross-sectional study. Instead, historical data on whether the participant had been diagnosed with asthma will be collected.

The cross-sectional study has several study groups based on the exposure (smoking behavior) status. Combinations of paired associations are as follows: smokers vs. never-smokers; smokers vs. ex-smokers; never-smokers vs. ex-smokers. Therefore, it bears some feature of a retrospective cohort study, specifically; it provides an opportunity to make comparisons between the groups. While calculating the required sample size, the investigators considered this opportunity as the most important one. In addition to calculating prevalence ratio of COPD for exposure statuses, the cross-sectional study will allow for assessment of prevalence of these conditions and other characteristics in different study groups.

Data to be collected

* Spirometry (FEV / FVC), bronchodilation test
* COPD assessment test (CAT) questionnaire,
* 6-minute walk test
* Electrocardiography
* High-resolution computed tomographic (HRCT) scan of the chest
* Blood pressure
* Body mass index (BMI)
* Smoking status and history
* Passive smoking status
* Occupational exposure
* Exposure to indoor biofuel pollution
* Patient-reported comorbidities
* Laboratory testing for: blood cholesterol level, HDL (high-density lipoprotein), LDL (low-density lipoproteins), triglycerides, C-reactive protein, fibrinogen, glucose, Hepatitis B and C IgM and IgG antigens and antibodies, liver enzymes (ALT and AST), and alpha-1-antitrypsine.

The investigators plan to recruit subjects by using the following mechanisms, namely, through social media, a network of medical referral sites (polyclinics and ambulatory centers), and from large corporations, i.e. with more than 500 employees.

Information about current smoking behavior and very detailed historic information on smoking behavior will be used to for adjustments during the data analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* ≥10 pack-year smoking history (for smokers and ex-smokers)
* less than 100 cigarettes in lifetime (for never-smokers)
* be able to provide informed consent

Exclusion Criteria:

* be pregnant
* has a fever (370C or higher) at the time of the visit and during the last two weeks preceding the visit
* be legally incapable
* chronic infectious and non-infectious lung disease except asthma (eg, pulmonary fibrosis, bronchiectasis, cystic fibrosis, tuberculosis, and others.)
* resection of at least one lobe (or performing procedures to reduce lung volume)
* any cancer and receiving a course of radiation and/or chemotherapy at the time of the visit;
* suspected lung cancer (presence of significant lung neoplasm)
* presence of metal in the chest
* ophthalmic surgery within the last 12 months prior to the visit
* myocardial infarction or other form of acute or chronic coronary insufficiency, cardiac arrhythmias diagnosed of at least 6 months prior to the visit
* myocardial infarction or other form of acute or chronic coronary insufficiency, cardiac arrhythmias with which an individual regularly receives medication
* Severely elevated blood pressure (equal to or greater than a systolic 180 or diastolic of 100)
* history of cerebrovascular accidents
* thoracic or abdominal surgery within the last 6 months
* contraindications to use salbutamol or its analogues
* CT scan or other research using ionizing radiation within the last 6 months

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is three groups of male and female residents of City of Almaty, the largest city in Kazakhstan, with a population of 1,7 million people, containing 9% of the country's total population aged 33-59. The first group is current smokers with more than 10 pack-year history of smoking. The second group is individuals who quitted smoking from one to five years ago and have more than 10 pack-year history of smoking. The third group is persons who has never smoked regularly, i.e. smoked less than 100 cigarettes in his or her lifetime.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Evidence of chronic obstructive pulmonary disease | up to 1 week
  airflow obstruction based on the fixed ratio of post-bronchodilator FEV1 /FVC < 0.70 criterion

SECONDARY OUTCOMES:
Airflow obstruction through lung function test | up to 1 week
  Items to be analyzed are pre/post bronchodilator FEV1, FVC, FEV1/FVC
COPD CT score | up to 2 weeks
  Semi-quantified measures performed by three CT scan readers to evaluate extent of emphysema, severity of bronchial dilatation, traction bronchiectasis, bronchial wall thickening, small airways disease
Results of 6-minute walking test | up to 1 week
COPD assessment test (CAT) score | up to 1 week
Comorbidities of COPD | up to 1 week
Presence of metabolic syndrome | up to 1 week
  Detection of metabolic syndrome based on the new International Diabetes Federation (IDF) definition that includes central obesity AND any two of the following factors: raised TG level; reduced HDL cholesterol; raised blood pressure; raised fasting plasma glucose
10 year risk of fatal CVD | up to 1 week
  Systematic Coronary Risk Evaluation (SCORE) based on the European High Risk SCORE Chart by gender, age, systolic blood pressure, total cholesterol and smoking status
Presence of an electrocardiogram abnormality | up to 1 week
  Detection of abnormality during the electrocardiogram

OTHER OUTCOMES:
Concentrations of total cholesterol, low density lipoprotein (LDL) cholesterol, HDL cholesterol, triglyceride (TG), glucose, liver enzymes (ALT and AST), C-reactive protein, fibrinogen, and alpha-1-antitrypsin | up to 1 week
  Serum laboratory testing for blood cholesterol level, HDL (high-density lipoprotein), LDL (low-density lipoproteins), triglycerides, C-reactive protein, fibrinogen, glucose, liver enzymes (ALT and AST), and alpha-1-antitrypsin
Number of Participants With Positive or Negative Results of Testing for Anti-HCV and HBsAG | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Almaz T Sharman, MD, PhD, Principal Investigator — Kazakhstan Academy of Preventive Medicine
Locations (1):
- Kazakhstan Academy of Preventive Medicine, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share all participant data except personally identifiable information. Data will be available to open-access after the completion of the study (after July 31, 2017). Access to study data, which is going to be located in our web site, will be granted by request.

REFERENCES:
- [Derived] Sharman A, Zhussupov B, Sharman D, Stambekova A, Yeraliyev S. Cross-Sectional Study of Chronic Obstructive Pulmonary Disease Prevalence Among Smokers, Ex-Smokers, and Never-Smokers in Almaty, Kazakhstan: Study Protocol. JMIR Res Protoc. 2017 Jul 25;6(7):e143. doi: 10.2196/resprot.7422. PMID 28743683